CLINICAL TRIAL: NCT03391869
Title: Randomized Phase III Trial of Local Consolidation Therapy (LCT) After Nivolumab and Ipilimumab for Immunotherapy-Naive Patients With Metastatic Non-Small Cell Lung Cancer (LONESTAR)
Brief Title: Nivolumab and Ipilimumab With or Without Local Consolidation Therapy in Treating Patients With Stage IV Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0311; NCI-2018-00825 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0311 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-01-02; First posted 2018-01-05 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Lung Adenocarcinoma; Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (ipilimumab, nivolumab) (Experimental): INDUCTION PHASE: Patients receive nivolumab IV over 90 minutes on days 1, 15, and 29, and ipilimumab IV over 60 minutes on day 1. Treatment repeats every 6 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  Patients receive nivolumab IV over 60 minutes on days 1, 15, and 29 and ipilimumab IV over 90 minutes on day 1. Courses repeat every 6 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab; Other: Quality-of-Life Assessment
- Arm B (ipilimumab, nivolumab, LCT) (Experimental): INDUCTION PHASE: Patients receive nivolumab IV over 90 minutes on days 1, 15, and 29, and ipilimumab IV over 60 minutes on day 1. Treatment repeats every 6 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  Patients receive LCT consisting of surgery and/or radiation 14 days after completion of Induction Phase. Patients then receive nivolumab and ipilimumab as in arm A beginning within 4 weeks after LCT. Courses repeat every 6 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Procedure: Local Consolidation Therapy; Biological: Nivolumab; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy
Procedure: Local Consolidation Therapy — Undergo radiation and/or surgery
  Other Names: LCT; Local Consolidative Therapy
  Arms: Arm B (ipilimumab, nivolumab, LCT)
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Undergo radiation
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Arm B (ipilimumab, nivolumab, LCT)
Procedure: Therapeutic Conventional Surgery — Undergo surgery
  Arms: Arm B (ipilimumab, nivolumab, LCT)

SUMMARY:
This phase III trial studies how well nivolumab and ipilimumab works with or without local consolidation therapy in treating patients with stage IV non-small cell lung cancer. Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Local consolidation therapy, such as surgery or radiation therapy, may improve survival outcomes in patients with non-small cell lung cancer. It is not yet known whether giving nivolumab and ipilimumab with local consolidation therapy works better than nivolumab and ipilimumab alone in treating patients with stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether local consolidative therapy (LCT; radiotherapy +/- surgical resection, radiofrequency ablation, or cryoablation for up to 3 lesions) followed by up to 2 years of treatment with ipilimumab (1mg/Kg every 6 weeks) and nivolumab (3 mg/Kg, every 2 weeks) prolongs overall survival (OS) compared with up to 2 years treatment with ipilimumab (1mg/Kg every 6 weeks) and nivolumab (3 mg/Kg, every 2 weeks) alone in metastatic or recurrent non-small cell lung cancer (NSCLC) patients with non-progressive disease after 12 weeks of treatment with ipilimumab (1mg/Kg every 6 weeks) and nivolumab (3 mg/Kg, every 2 weeks).

II. Determine whether LCT followed by up to 2 years of treatment with ipilimumab (1mg/Kg every 6 weeks) and nivolumab (3 mg/Kg, every 2 weeks) prolongs overall survival compared with up to 2 years of treatment with ipilimumab (1mg/Kg every 6 weeks) and nivolumab (3 mg/Kg, every 2 weeks) alone in the subgroup of patients with oligometastatic NSCLC (up to 3 metastases) with non-progressive disease after 12 weeks of treatment with ipilimumab (1mg/Kg every 6 weeks) and nivolumab (3 mg/Kg, every 2 weeks).

SECONDARY OBJECTIVES:

I. To determine if there is a progression free survival (PFS) difference in the overall group and the oligometastatic group in patients that receive LCT + ipilimumab/nivolumab vs. ipilimumab/nivolumab alone.

II. To determine whether there is a PFS and (overall survival) OS difference in patients that undergo complete vs. non-complete LCT after 12 weeks of induction treatment with ipilimumab (1mg/Kg every 6 weeks) and nivolumab (3 mg/Kg, every 2 weeks).

III. To determine whether LCT improves time to progression of non-irradiated lesions (TTP-NIL) and time to appearance of new metastases (TANM) in the overall study population and the oligometastatic subgroup.

IV. To determine whether LCT improves the time to progression of target vs. non-target lesions in the overall study population and the oligometastatic subgroup.

V. To assess whether LCT prolongs PFS and OS in squamous histology and non-squamous histologies.

VI. To assess the safety and tolerability of nivolumab and ipilimumab with or without LCT.

VII. To assess quality of life patient reported outcomes in patients treated with nivolumab and ipilimumab with or without LCT.

VIII To explore the association of baseline genomic and gene expression profiles (from tumor, germline deoxyribonucleic acid [DNA], and cell free [cf] DNA) with clinical benefit and toxicities in patients treated with nivolumab and ipilimumab with or without LCT.

IX. To explore the association of baseline immune profiles (from tumor and blood) with clinical benefit and toxicities in patients treated with nivolumab and ipilimumab with or without LCT.

EXPLORATORY OBJECTIVE:

I. To identify novel prognostic and predictive markers present at diagnosis, and to determine modulation of markers by induction immunotherapy in order to inform future translational studies.

OUTLINE:

INDUCTION PHASE: Patients receive nivolumab intravenously (IV) over 90 minutes on days 1, 15, and 29, and ipilimumab IV over 60 minutes on day 1. Treatment repeats every 6 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity.

Patients with non-progressive disease after completion of Induction Phase are randomized to 1 of 2 arms.

ARM A: Patients receive nivolumab IV over 60 minutes on days 1, 15, and 29 and ipilimumab IV over 90 minutes on day 1. Courses repeat every 6 weeks for 2 years in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive LCT consisting of surgery and/or radiation 14 days after completion of Induction Phase. Patients then receive nivolumab and ipilimumab as in arm A beginning within 4 weeks after LCT. Courses repeat every 6 weeks for 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 8 weeks and then every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer; if a diagnostic biopsy is available, a pre-treatment biopsy is not required. Patients with a suspected lung cancer may be consented, but pathology must be confirmed prior to initiating treatment on study. Neuroendocrine carcinomas (e.g. small cell lung cancer [SCLC], carcinoid tumors) are not eligible. Carcinomas with neuroendocrine differentiation are eligible.
* Stage IV (according to the American Joint Committee on Cancer [AJCC] 8th edition) measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Signed and dated written or remote informed consent prior to admission to the study in accordance with International Conference on Harmonization-Good Clinical Practice (ICH-GCP) guidelines and to the local legislation.
* For lung adenocarcinoma patients, patients must not harbor any EGFR sensitizing or ALK fusion where there are standard care therapy options available. For patients with histologies other than adenocarcinoma, EGFR and ALK status is not required. Adenocarcinoma patients may be consented prior to the EGFR and ALK status being known, but EGFR and ALK status must be determined prior to initiating therapy. EGFR and ALK status may be determined using either tumor- or plasma-based, Clinical Laboratory Improvement Amendments (CLIA)-certified assays. For patients with non-small cell lung cancer (NSCLC), not otherwise specified (NOS), EGFR/ALK testing is not required, as the frequency of alterations is exceedingly rare in this histology. Also, note that patients with ROS1/RET alterations can be enrolled, as tyrosine kinase inhibitor such as crizotinib aren't established as first line therapy for patients with these alterations.
* One prior line of chemotherapy and/or targeted agents for metastatic disease are permitted. This chemotherapy can include maintenance therapy, as long as it was given in the front line setting. In addition, prior antiangiogenic therapy (e.g. bevacizumab) is permitted if used as frontline treatment.

Patients must have organ and marrow function as defined below:

* Performance status of 0 or 1 if using Eastern Cooperative Oncology Group (ECOG)/Zubrod.
* Screening laboratory values must meet the following criteria and should be obtained within 14 days prior to treatment initiation
* White blood cell (WBC ) >= 2000/uL
* Neutrophils >= 1500/uL (obtained within 14 days prior to randomization/registration)
* Platelets >= 100 x 10^3/uL (obtained within 14 days prior to randomization/registration)
* Hemoglobin > 9.0 g/dL (obtained within 14 days prior to randomization/registration)
* Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or creatinine clearance (CrCl) ≥ 50 mL (if using the Cockcroft-Gault formula)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 3 x ULN (obtained within 14 days prior to randomization/registration)
* Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert syndrome, who can have total bilirubin < 3.0 mg/dL) (obtained within 14 days prior to randomization/registration)
* Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. Appropriate methods of contraception are as follows. Women will be instructed to adhere to contraception for a period of 26 weeks after the last dose of investigational product. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 35 weeks after the last week of nivolumab/ipilimumab (nivo/ipi). Note: WOCBP is defined as any female who has experienced menarche and who has not yet undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented negative serum or urine test.
* Women of childbearing potential must have a negative serum or urine pregnancy test within 48 hours prior to the start of nivolumab.
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 35 weeks after the last dose of investigational product. Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile) as well as azoospermic men do not require contraception.
* Subjects with brain metastases are eligible if metastases are adequately treated and subjects are neurologically stable (except for residual signs or symptoms related to the central nervous system [CNS] treatment) for at least 2 weeks prior to the first dose of nivolumab. In addition, subjects must be either off corticosteroids, or on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent) for at least 2 weeks prior to the first dose of nivolumab. Patients with asymptomatic, small (e.g. =< 1 cm) brain metastases are 1) eligible provided that the patient is off corticosteroids, or on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent) for at least 2 weeks prior to the first dose of nivolumab
* For cohort 1 subjects may receive radiotherapy for symptomatic metastases prior to enrollment provided that there is at least one other non-irradiated lesion amenable to LCT at the time of enrollment. When feasible, stereotactic body radiation therapy (SBRT) or other hypofractionated techniques are strongly encouraged.

Inclusion Criteria In Cohort 2:

* Patients must have disease progression per imaging radiologic studies prior to randomization in LONESTAR study (during induction phase)
* Patient in this cohort must start therapy with platinum doublet and immune checkpoint inhibitor therapy no longer than 6 weeks after their last day of immune checkpoint inhibitor therapy
* Patients must have organ and marrow function as defined below:

Performance Status of 0 or 1 if using ECOG/Zubrod. Screening laboratory values must meet the following criteria and should be obtained within 14 days prior to treatment initiation

WBC ≥ 2000/μL Neutrophils ≥ 1500/μL Platelets ≥ 100 x103/μL Hemoglobin > 9.0 g/dL

Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 50 mL (if using the Cockcroft-Gault formula below):

AST/ALT ≤ 3 x ULN Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)

* Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. Appropriate methods of contraception are as follows. Women will be instructed to adhere to contraception for a period of 26 weeks after the last dose of investigational product. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 35 weeks after the last week of nivo/ipi. Note: WOCBP is defined as any female who has experienced menarche and who has not yet undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented negative serum or urine test.
* Women of childbearing potential must have a negative serum or urine pregnancy test within 48 hours prior to the start of therapy.
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 35 weeks after the last dose of investigational product Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception.Subjects with brain metastases are eligible if metastases are adequately treated (exception of ≤1 cm asymptomatic brain metastases, as specified below) and subjects are neurologically stable (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to the first dose of nivolumab. In addition, subjects must be either off corticosteroids, or on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent) for at least 2 weeks prior to the first dose of nivolumab. In addition, subjects must be either off corticosteroids or on stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent) for at least 2 weeks prior to the first dose of nivolumab. Patients with asymptomatic, small (e.g. ≤1 cm) brain metastases are eligible and do not require prior local therapy for eligibility, provided that the patient is off corticosteroids, or on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent) for at least 2 weeks prior to the first dose of nivolumab.
* Participants enrolled in the cohort 2 must be willing to undergo tumor biopsy prior to the initiation of therapy with immune checkpoint inhibitor and platinum doublet therapy and on treatment biopsies. In cases when such a biopsy is clinically unsafe to perform, archival (meaning obtained at earlier times) tumor biopsies may be accepted the discretion of the study PI.
* For cohort 2 subjects may receive radiotherapy for symptomatic metastases at the time of their progression prior to enrollment to cohort 2

Exclusion Criteria:

* Systemic immunotherapy for metastatic NSCLC. Immunotherapy agents include, but are not limited to, agents targeting the PD1/PD-L1 axis (e.g. nivolumab, pembrolizumab, atezolizumab, durvalumab) or CTLA-4 (ipilimumab, tremelimumab) pathways.
* Any approved anti-cancer therapy, including chemotherapy, or hormonal therapy within 3 weeks prior to the initiation of study treatment. The following exceptions are allowed: hormone-replacement therapy or oral contraceptives
* Women must not be breastfeeding.
* Patients excluded with any prior treatment of pneumonitis requiring corticosteroids within 60 days prior to the first dose of nivolumab
* Unwillingness or inability to follow the procedures required in the protocol.
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
* Prior malignancy active within the previous 2 years. Patients with locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast with local control measures (surgery, radiation) are eligible.
* Patients should be excluded if they have an active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration (i.e. disease-modifying antirheumatic drugs). Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Note that subjects are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if >10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g. contrast dye allergy) or for treatment of non-autoimmune conditions (e.g. delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
* As there is potential for hepatic toxicity with nivolumab or nivolumab/ipilimumab combinations, drugs with a predisposition to hepatoxicity should be used with caution.
* Patients should be excluded if they are known to be positive for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.
* Patients should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* History of allergy to study drug components.
* History of severe hypersensitivity reaction to any monoclonal antibody.
* Prisoners or subjects who are involuntarily incarcerated.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (infection disease) illness.
* Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule.
* Any condition that, in the opinion of the investigator, would interfere with the study treatment or interpretation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) in overall population | Up to 1 year after completion of study treatment
  The type I error of 0.10 for the entire study is divided in half (0.10/2 = 0.05) allowing for a Type I error of 0.05 for each of the efficacy endpoints.
OS in oligometastatic subgroup | Up to 1 year after completion of study treatment
  The assessment for the subpopulation of patients with oligometastatic disease will be conducted only if the finding in the total population is found to be non-significant. The type I error of 0.10 for the entire study is divided in half (0.10/2 = 0.05) allowing for a Type I error of 0.05 for each of the efficacy endpoints described above.

CONTACTS AND LOCATIONS:
Overall Officials: John V Heymach, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - MD Anderson in The Woodlands, Conroe, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas

REFERENCES:
- [Derived] Altan M, Li R, Li Z, Chen R, Sheshadri A, Tran HT, Little L, Baguley J, Sinson J, Vokes N, Gandhi S, Antonoff MB, Swisher SG, Lizee G, Reuben A, Heymach JV, Zhang J. High peripheral T cell diversity is associated with lower risk of toxicity and superior response to dual immune checkpoint inhibitor therapy in patients with metastatic NSCLC. J Immunother Cancer. 2024 Dec 25;12(12):e008950. doi: 10.1136/jitc-2024-008950. PMID 39721752
- [Derived] Altan M, Li QZ, Wang Q, Vokes NI, Sheshadri A, Gao J, Zhu C, Tran HT, Gandhi S, Antonoff MB, Swisher S, Wang J, Byers LA, Abdel-Wahab N, Franco-Vega MC, Wang Y, Lee JJ, Zhang J, Heymach JV. Distinct patterns of auto-reactive antibodies associated with organ-specific immune-related adverse events. Front Immunol. 2023 Dec 12;14:1322818. doi: 10.3389/fimmu.2023.1322818. eCollection 2023. PMID 38152395
- See also: MD Anderson Cancer Center — http://www.mdanderson.org